CLINICAL TRIAL: NCT06758362
Title: Comparison of Online EMDR Therapy and CBT for PTSD Symptoms Following the Kahramanmaraş Earthquakes: a Randomized Controlled triaL
Brief Title: EMDR vs. CBT for PTSD
Acronym: EARTH-PTSD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Collaborators: Uskudar University (Other); Beykoz University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Assistant Professor in Psychology Department, Principle investigator, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nisantasi U
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: Post-Traumatic Stress Disorder (PTSD); Eye Movement Desensitization and Reprocessing (EMDR); Cognitive Behavioral Therapy (CBT); Earthquake Survivors; Kahramanmaraş Earthquakes
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Model Description:
  This study follows an Interventional, Parallel-Group, Open-Label, Randomized Controlled Trial (RCT) design to compare the effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) and Cognitive Behavioral Therapy (CBT) in reducing post-traumatic stress disorder (PTSD) symptoms among survivors of the 2023 Kahramanmaraş earthquakes.
  Study Design Details:
  Interventional Model: Parallel Assignment
  Participants will be randomly assigned to one of three distinct groups:
  EMDR Therapy Group: Weekly 50-minute sessions for 12 weeks CBT Therapy Group: Weekly 50-minute sessions for 12 weeks Control Group: No therapeutic intervention during the study period Masking: None (Open-Label) Participants and therapists will know the assigned intervention group. Purpose: Treatment To compare the therapeutic outcomes of EMDR and CBT in alleviating PTSD symptoms.
  Intervention Delivery: Online, one-on-one therapy sessions using Microsoft Teams.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- EMDR Therapy Group (Active Comparator): Arm Description: Interventional Study
  Participants in the EMDR Therapy Group will receive Eye Movement Desensitization and Reprocessing (EMDR) therapy, a structured, evidence-based psychotherapy approach specifically designed to alleviate symptoms of post-traumatic stress disorder (PTSD).
  Intervention Details:
  Weekly 50-minute individual online therapy sessions conducted via Microsoft Teams.
  A total of 12 sessions delivered over 12 weeks. Sessions will follow standard EMDR protocols, including assessment, preparation, desensitization, installation, and re-evaluation phases.
  Therapists:
  Sessions will be conducted by trained EMDR therapists: Dr. Eda Yılmazer. The primary goal is to assess the effectiveness of EMDR therapy in reducing PTSD symptoms among earthquake survivors. Therapy adherence and quality will be monitored throughout the intervention period.
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)
- CBT Interventional Group (Active Comparator): Arm Description:
  Participants in the CBT Therapy Group will receive Cognitive Behavioral Therapy (CBT), a well-established, evidence-based psychotherapy approach aimed at reducing symptoms of post-traumatic stress disorder (PTSD) by addressing maladaptive thought patterns and behaviors.
  Intervention Details:
  Weekly 50-minute individual online therapy sessions conducted via Microsoft Teams.
  A total of 12 sessions delivered over 12 weeks. Sessions will follow standard CBT protocols, focusing on identifying and challenging negative thought patterns, developing coping strategies, and gradually reducing trauma-related distress.
  Therapists:
  Sessions will be conducted by trained CBT therapists: Dr. Selami Varol Ülker and Dr. Metin Çınaroğlu.
  The primary goal is to assess the effectiveness of CBT in reducing PTSD symptoms among earthquake survivors. Therapy adherence and quality will be monitored throughout the intervention period.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)
- Control Group (No Intervention): Arm Description:
  Participants in the Control Group will not receive any therapeutic intervention during the study period. They will serve as a comparison group to evaluate the effectiveness of Eye Movement Desensitization and Reprocessing (EMDR) and Cognitive Behavioral Therapy (CBT) in reducing post-traumatic stress disorder (PTSD) symptoms.
  Intervention Details:
  No active therapy sessions will be provided. Participants will continue with their usual daily routines without any specific psychological intervention.
  Assessments:
  Participants will undergo the same PTSD symptom assessments as the intervention groups at four time points:
  Before the study begins (Baseline) After the 6th week (Midpoint) After the 12th week (End of study) This group will provide essential comparative data to measure the relative effectiveness of EMDR and CBT in alleviating PTSD symptoms among earthquake survivors.

INTERVENTIONS:
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — A structured psychotherapy approach focused on reducing PTSD symptoms through guided eye movements and trauma processing.
  Arms: EMDR Therapy Group
Behavioral: Cognitive Behavioral Therapy (CBT) — A psychotherapy approach focused on identifying and modifying maladaptive thought patterns and behaviors to reduce PTSD symptoms.
  Arms: CBT Interventional Group

SUMMARY:
This study compares two evidence-based therapies, Eye Movement Desensitization and Reprocessing (EMDR) and Cognitive Behavioral Therapy (CBT), in reducing symptoms of post-traumatic stress disorder (PTSD) among adults affected by the 2023 Kahramanmaraş earthquakes in Türkiye. A total of 89 participants diagnosed with PTSD were randomly assigned to one of three groups: EMDR therapy, CBT therapy, or a no-treatment control group. Each participant in the treatment groups received 12 weekly, one-on-one, 50-minute therapy sessions delivered remotely via a secure online platform. PTSD and related symptoms (depression, anxiety, and emotion dysregulation) were assessed at three time points: before therapy (T1), after the 6th session (T2), and after the 12th session (T3). This study aims to evaluate which therapy yields stronger improvements in PTSD and related psychological outcomes when delivered remotely in a disaster-affected population.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to compare the effectiveness of two trauma-focused psychotherapeutic interventions-Eye Movement Desensitization and Reprocessing (EMDR) and Cognitive Behavioral Therapy (CBT)-in alleviating post-traumatic stress disorder (PTSD) symptoms among adult survivors of the 2023 Kahramanmaraş earthquakes in Türkiye. These earthquakes caused large-scale devastation across 11 cities and resulted in significant psychological distress, including high rates of PTSD.

Study Objectives:

The primary objective was to determine whether EMDR or CBT is more effective in reducing PTSD symptoms, as measured by the PTSD Checklist for DSM-5 (PCL-5). Secondary objectives included examining changes in depressive symptoms, anxiety, and emotion regulation difficulties over the course of treatment.

Study Design:

This was an open-label, three-arm, randomized controlled trial. A total of 89 adult participants (aged 18-65) who met DSM-5 criteria for PTSD (based on clinical interview and PCL-5 scores) were randomly assigned to one of three groups:

EMDR Therapy Group (n = 30) CBT Therapy Group (n = 30) No-Treatment Control Group (n = 29)

Intervention Delivery:

Each participant in the therapy arms received 12 weekly, 50-minute, one-on-one sessions delivered remotely via Microsoft Teams. The control group received no intervention during the study period but underwent the same assessments.

Intervention Details:

EMDR Therapy: Delivered by certified EMDR therapists using the standard 8-phase protocol, adapted for remote delivery with visual and tactile bilateral stimulation.

CBT Therapy: Delivered by certified CBT therapists following trauma-focused CBT protocols, including psychoeducation, cognitive restructuring, and behavioral activation.

Outcome Measures:

Primary Outcome: PTSD symptoms assessed using the PCL-5 at three time points: baseline (T1), after the 6th session (T2), and after the 12th session (T3).

Secondary Outcomes: Depression (BDI-II), anxiety (BAI), and emotion regulation (DERS).

Supervision and Quality Control:

All therapists were supervised weekly by a senior psychiatrist. A fidelity monitoring committee reviewed random session recordings for quality control.

Ethical Considerations:

The study was approved by the Üsküdar University Non-Invasive Research Ethics Committee (Approval No: 61351342/020-316). Informed consent and publication consent were obtained from all participants.

Timeline:

Recruitment: January-March 2025 Intervention: April-June 2025 Follow-Up: A separate long-term follow-up is planned and will be reported in a subsequent study.

Expected Outcomes:

The study aims to provide empirical evidence on the feasibility and effectiveness of online EMDR and CBT for PTSD in disaster-affected populations, informing scalable intervention strategies for future post-disaster mental health services.

ELIGIBILITY:
Eligibility Criteria

* Minimum Age: 18 Years
* Maximum Age: 65 Years
* Sex: All
* Gender Based: No
* Accepts Healthy Volunteers: No

Inclusion Criteria:

* Adults aged 18-65 years.
* Diagnosed with Post-Traumatic Stress Disorder (PTSD) based on the PTSD ---Checklist for DSM-5 (PCL-5) and Clinician-Administered PTSD Scale (CAPS-5).
* Resided in the Kahramanmaraş earthquake-affected region during the disaster.
* No current psychiatric medication or ongoing psychotherapy.
* No history of psychiatric disorders that may interfere with PTSD treatment (e.g., bipolar disorder, schizophrenia, substance-related disorders).
* Ability to attend weekly, one-on-one, 50-minute online therapy sessions for 24 weeks.
* Provided written informed consent and psychiatric clearance for study participation.

Exclusion Criteria:

* Individuals currently undergoing psychotherapy or using psychiatric medications.
* Diagnosis of bipolar disorder, schizophrenia, substance-related disorders, or other psychiatric conditions that may interfere with treatment.
* Inability to commit to 24 weeks of therapy sessions or attend sessions online.
* Severe cognitive impairment preventing participation in therapy.
* Failure to provide written informed consent or psychiatric clearance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Reduction in PTSD Symptom Severity Measured by the PTSD Checklist for DSM-5 (PCL-5) | Time Frame: Baseline (Before therapy begins) After the 6th session (Mid-therapy, approximately 6 weeks) After the 12th session (Post-therapy, approximately 12 weeks) Six months post-therapy
  The primary outcome will measure changes in PTSD symptom severity using the PTSD Checklist for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (PCL-5), a validated self-report questionnaire designed to assess PTSD symptom severity based on DSM-5 criteria.
  Scale Details:
  Minimum Score: 0 Maximum Score: 80 Score Interpretation: Higher scores indicate worse PTSD symptom severity, while lower scores indicate improvement.
  Assessment Time Points:
  Baseline (Before therapy begins) After the 6th session (Mid-therapy, approximately 6 weeks) After the 12th session (Post-therapy, approximately 12 weeks) The analysis will focus on changes in total PCL-5 scores across these time points to compare the effectiveness of EMDR and CBT therapies in addressing PTSD symptoms relative to the Control Group.

SECONDARY OUTCOMES:
Change in depressive symptoms as measured by the Beck Depression Inventory-II (BDI-II) | Baseline (pre-treatment), after session 6 (mid-treatment), and after session 12 (post-treatment)
  This secondary outcome will measure changes in depressive symptom severity using the Beck Depression Inventory-II (BDI-II), a widely used 21-item self-report questionnaire designed to assess cognitive, affective, and somatic symptoms of depression over the previous two weeks.
  Scale Details:
  Minimum Score: 0 Maximum Score: 63 Score Interpretation: Higher scores indicate more severe depressive symptoms; lower scores indicate clinical improvement.
  Assessment Time Points:
  Baseline (Before therapy begins) After the 6th session (Mid-therapy, approximately 6 weeks) After the 12th session (Post-therapy, approximately 12 weeks) The analysis will examine changes in total BDI-II scores over time to evaluate and compare the effects of EMDR and CBT on depression in earthquake survivors.
Change in anxiety symptoms as measured by the Beck Anxiety Inventory (BAI) | Baseline (pre-treatment), after session 6 (mid-treatment), and after session 12 (post-treatment)
  This secondary outcome will assess changes in anxiety symptoms using the Beck Anxiety Inventory (BAI), a 21-item self-report measure that evaluates the intensity of physiological and subjective symptoms of anxiety experienced during the past week.
  Scale Details:
  Minimum Score: 0 Maximum Score: 63 Score Interpretation: Higher scores indicate greater anxiety severity; lower scores reflect symptom reduction.
  Assessment Time Points:
  Baseline (Before therapy begins) After the 6th session (Mid-therapy, approximately 6 weeks) After the 12th session (Post-therapy, approximately 12 weeks) The analysis will focus on changes in total BAI scores across these time points to compare the therapeutic outcomes of EMDR and CBT for anxiety symptoms.
Change in emotion regulation difficulties as measured by the Difficulties in Emotion Regulation Scale (DERS) | Baseline (pre-treatment), after session 6 (mid-treatment), and after session 12 (post-treatment)
  This secondary outcome will measure changes in emotion regulation capacity using the Difficulties in Emotion Regulation Scale (DERS), a 36-item self-report instrument designed to assess individuals' typical levels of emotion dysregulation across six domains, including impulse control and emotional awareness.
  Scale Details:
  Minimum Score: 36 Maximum Score: 180 Score Interpretation: Higher scores indicate greater difficulties in emotion regulation; lower scores indicate better emotion regulation abilities.
  Assessment Time Points:
  Baseline (Before therapy begins) After the 6th session (Mid-therapy, approximately 6 weeks) After the 12th session (Post-therapy, approximately 12 weeks) The analysis will evaluate changes in total DERS scores to determine whether EMDR and CBT have differential effects on emotional regulation skills in the context of trauma recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Gökben Hızlı Sayar, Prof, Study Chair — Üsküdar University
Locations (1):
- Nişantaşı University, Istanbul, Maslak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Description:
  De-identified Individual Participant Data (IPD) will be shared with other researchers upon reasonable request to promote transparency, reproducibility, and further scientific exploration. The shared data will include:
  De-identified participant-level data for primary and secondary outcome measures Study protocol Statistical analysis plan
  Data Availability Timeline:
  Data will be made available 12 months after the publication of the primary results and will remain accessible for 5 years.
  Access Criteria:
  Researchers must submit a formal request outlining the purpose of data use, and approval will be granted by the principal investigators. Data will be shared via a secure data-sharing platform, ensuring compliance with ethical guidelines and data protection regulations.
  Contact Information:
  Requests for IPD access should be directed to the Principal Investigator, Dr. Metin Çınaroğlu, at metincinaroglu@gmail.com.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Time Frame:
  Start Date: 12 months after the publication of the primary study results End Date: 5 years after the start date
Access Criteria: Who Can Access:
  Researchers affiliated with academic institutions, non-profit organizations, or governmental research agencies who are conducting research aligned with the study's goals and objectives.
  What Can Be Accessed:
  De-identified Individual Participant Data (IPD) for all primary and secondary outcome measures.
  Supporting study documents, including the study protocol, statistical analysis plan, and informed consent forms (excluding participant identifiers).
  How to Access:
  Interested researchers must submit a formal written request to the Principal Investigator, including:
  A detailed research proposal outlining the purpose and scope of their study. Evidence of ethical approval for their research project from an accredited ethics board.
  Approved requests will be granted access to the data through a secure data-sharing platform under a data use agreement (DUA) that ensures compliance with ethical guidelines and data protection standards.